CLINICAL TRIAL: NCT05734807
Title: A Multicenter, Randomized, Controlled Phase IIa Study to Evaluate the Antiviral Activity and Safety of HH-003 in Nucleos(t)Ide Analogues-treated Chronic Hepatitis B Subjects With Low-Level Viremia
Brief Title: A Study to Evaluate the Antiviral Activity and Safety of HH-003 in Chronic Hepatitis B Subjects With Low-level Viremia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HH003-203
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic HBV Infection
MeSH Terms: interventions — Nucleosides

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NrtIs (Active Comparator)
  Interventions: Drug: Nucleoside/nucleotide reverse transcriptase inhibitors (NrtIs)
- HH-003+NrtIs (Experimental)
  Interventions: Drug: HH-003 and NrtIs
- HH-003+NrtIs+PEG-IFN-α (Experimental)
  Interventions: Drug: HH-003, NrtIs and PEG-IFN-α

INTERVENTIONS:
Drug: Nucleoside/nucleotide reverse transcriptase inhibitors (NrtIs) — Subjects will receive NrtIs therapy for 24 weeks.
  Arms: NrtIs
Drug: HH-003 and NrtIs — Subjects will receive HH-003 20 mg/kg intravenously Q2W and NrtIs therapy for 24 weeks.
  Arms: HH-003+NrtIs
Drug: HH-003, NrtIs and PEG-IFN-α — Subjects will receive HH-003 20 mg/kg intravenously Q2W, NrtIs therapy and PEG-IFN-α 180μg SC QW for 24 weeks.
  Arms: HH-003+NrtIs+PEG-IFN-α

SUMMARY:
This is a multicenter, randomized, controlled Phase IIa study of HH-003 to evaluate the antiviral activity and safety in nucleos(t)ide analogues-treated chronic hepatitis B subjects with low-level viremia. HH-003 is a human monoclonal antibody targeting the pre-S1 domain of the HBV large envelope protein. It blocks engagement of preS1 with sodium taurocholate co-transporting polypeptide (NTCP), the cellular receptor for HBV.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form;
* Male or female aged from 18 to 60 years (inclusively);
* 18 kg/m^2≤BMI≤30 kg/m^2, body weight≥50 kg for men and ≥45 kg for women;
* Subjects who have chronic HBV infection greater than or equal to 6 months at screening;
* 10 IU/mL≤HBsAg≤3000 IU/mL; HBV DNA≤2000 IU/mL; ALT≤3×ULN;
* Subjects who have been on nucleoside reverse transcriptase inhibitors therapy for more than 1 year prior to screening.

Exclusion Criteria:

* Females who are pregnant or lactating at screening;
* History of alcoholic liver disease, moderate fatty liver, autoimmune liver disease, other hereditary liver disease, drug-induced liver disease or other clinically significant chronic liver disease induced by non-HBV infection;
* History of cirrhosis at any time prior to or at time of screening, or having progressive liver fibrosis at screening ;
* History or evidence of hepatocellular carcinoma at any time prior to or at time of screening;
* Exclusionary laboratory results at screening: total bilirubin >2xULN or direct bilirubin >1.5xULN，hemoglobin <120 g/L for males or <110 g/L ro females，platelets count<100,000/mm^3 (100×10^9/L), and absolute neutrophils count <1,500/mm^3 (1.5×10^9/L).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with HBV DNA negativation | Week 24
Changes from baseline in serum HBsAg | From treatment start up to Week 48

SECONDARY OUTCOMES:
Percentage of subjects achieving maintained virologic response (MVR) | From treatment start up to 48 weeks
Duration of MVR | From treatment start up to 48 weeks
Percentage of subjects with ALT normalization | From treatment start up to 48 weeks
Changes from baseline in serum HBeAg in subjects with positive HBeAg | From treatment start up to 48 weeks

CONTACTS AND LOCATIONS:
Locations (8):
- China (8):
  - Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou, Fujian
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Sixth Peoples Hospital Of Zhengzhou, Zhengzhou, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shandong Public Health Clinical Center, Jinan, Shandong